CLINICAL TRIAL: NCT07329790
Title: Indian National Study to Assess Incidence and Severity of Post-ERCP Pancreatitis After Following SOP
Acronym: INSPIRE
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterology, Asian Institute of Gastroenterology, India
Other Study IDs: INSPIRE
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: ERCP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rectal NSAID Prophylaxis: Participants who receive a single dose of rectal indomethacin or diclofenac (100 mg suppository) as part of routine clinical practice. The dose is given 30 minutes before ERCP, or immediately after the procedure if the pre-procedure dose was missed.
- Pancreatic Duct Stent Placement: Participants in whom the pancreatic duct is accessed during ERCP and a small plastic prophylactic pancreatic duct stent is placed as part of standard care. The stent is temporary and is expected to pass naturally or be removed within 14 days

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an indispensable therapeutic procedure in the management of a wide spectrum of pancreaticobiliary disorders, including choledocholithiasis, benign and malignant biliary strictures, pancreatic ductal obstructions, and postoperative bile leaks. The procedure has revolutionized the management of these conditions, often obviating the need for surgery. However, despite its therapeutic efficacy, ERCP carries a significant risk of procedure-related adverse events, of which post-ERCP pancreatitis (PEP) is the most common and clinically important complication.

The reported incidence of PEP in prospective multicenter studies ranges from 7 % to 10 % in unselected populations, and may increase to 15 % or higher in high-risk subsets such as patients with difficult cannulation, sphincter of Oddi dysfunction, or a prior history of pancreatitis or PEP. Although the majority of cases are mild and self-limited, a small but important proportion (approximately 10-15 %) progress to moderate or severe disease, resulting in prolonged hospitalization, increased cost, and occasionally mortality.

Over the past two decades, extensive research has improved our understanding of PEP pathogenesis and risk stratification. Several patient-related (younger age, female sex, prior PEP or pancreatitis, sphincter of Oddi dysfunction, asymptomatic choledocholithiasis) and procedure-related (difficult cannulation, pancreatic duct contrast injection or guidewire passage, pancreatic sphincterotomy, endoscopic papillary balloon dilation) predictors have been identified.

ELIGIBILITY:
Inclusion Criteria:

Consecutive ERCPs during the enrollment window.

* Males and females between 18 and 75 years of age who ca comprehend instructions, follow study procedures, willing to sign an informed consent form and have a clinical indication to undergo a ERCP.
* Patients undergoing ERCP for therapeutic indications
* Patients with intact papilla

Exclusion Criteria:

* patient undergoing ERCP for diagnostic indications
* Acute pancreatitis
* Previous sphincterotomy
* Altered anatomy, defined as anatomical variations in which bile and/or pancreatic secretion donot enter the duodenum by way of the ampulla of Vater
* Pregnancy
* Signs of Congestive heart failure, such as pitting edema or a NYHA classification greater than class II heart failure.
* Respiratory insufficiency (pO2 < 60 mmHg or saturation < 90% despite FiO2 of 30% or requiring mechanical ventilation).
* Severe liver disease (cirrhosis and ascites)
* Contraindication for rectal indomethacin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2366
Sampling Method: Probability Sample
Enrollment: 2366 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-ERCP pancreatitis (PEP), defined as | 30 days
  * New or worsened abdominal pain after ERCP with serum amylase or lipase ≥3 × the upper limit of normal measured ≥24 hours post-procedure,
  * Accompanied by hospitalization or prolongation of hospital stay attributable to pancreatitis.

SECONDARY OUTCOMES:
Severity of PEP | 30 days
  Mild, moderate, or severe according to the Revised Atlanta Classification (based on organ failure and duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: MD NITIN JAGTAP, MD,DM, Principal Investigator — Asian Institute Of Gastroenterology Private Limited

IPD SHARING:
Plan to Share IPD: No